CLINICAL TRIAL: NCT01989143
Title: A Phase 1, Randomzied, Double-blind, Third-party Open Placebo-controlled, Dose Escalating Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single Intravenous And Multiple Subcutaneous And Intravenous Doses Of Pf-06480605 In Healthy Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Intravenous and Multiple Subcutaneous and Intravenous Doses of PF-06480605 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telavant, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: B7541001
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Phase 1; Randomized; Double-blind; Placebo-controlled; Dose escalating; Single and Multiple doses; Safety; Tolerability; PK/PD; PF-06480605

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SAD Cohorts 1-8 Experimental Arm (Experimental)
  Interventions: Drug: PF-06480605
- SAD Cohorts 1-8 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD Cohorts 9-11 Experimental Arm (Experimental)
  Interventions: Drug: PF-06480605
- MAD Cohorts 9-11 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- MAD Cohort 12 Experimental Arm (Experimental)
  Interventions: Drug: PF-06480605
- MAD Cohort 12 Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06480605 — Subjects will receive single intravenous doses of 1, 3, 10, 30, 100, 300, 600 or 800 mg of PF-06480605 solution in a dose escalation format.
  Arms: SAD Cohorts 1-8 Experimental Arm
Drug: Placebo — Subjects will receive single intravenous doses of PF-06480605 matching placebo solution in a dose escalation format.
  Arms: SAD Cohorts 1-8 Placebo Arm
Drug: PF-06480605 — Subjects will receive three subcutaneous doses of 30, 100, or 300 mg of PF-06480605 solution in a dose escalation format of one dose every 2 weeks (q2wk).
  Arms: MAD Cohorts 9-11 Experimental Arm
Drug: Placebo — Subjects will receive three subcutaneous doses of PF-06480605 matching placebo solution in a dose escalation format of one dose every 2 weeks (q2wk).
  Arms: MAD Cohorts 9-11 Placebo Arm
Drug: PF-06480605 — Subjects will receive three intravenous doses of 500 mg of PF-06480605 solution in a dose escalation format of one dose every 2 weeks (q2wk).
  Arms: MAD Cohort 12 Experimental Arm
Drug: Placebo — Subjects will receive three intravenous doses of PF-06480605 matching placebo solution in a dose escalation format of one dose every 2 weeks (q2wk).
  Arms: MAD Cohort 12 Placebo Arm

SUMMARY:
This single and multiple ascending dose study is a first in human assessment of PF-06480605. The goal is to study the safety, tolerability, pharmacokinetics and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Female subjects of non childbearing potential must meet at least one of the following criteria:

  1. Achieved postmenopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females;
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
* X-ray with no evidence of current, active TB or previous inactive TB, general infections, heart failure, malignancy, or other clinically significant abnormalities taken at Screening or within 3 months prior to Day 1 and read by a qualified radiologist.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with a history of or current positive results for any of the following serological tests: Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), anti Hepatitis C antibody (HCV Ab) or human immunodeficiency virus (HIV).
* Subjects with a history of autoimmune disorders.
* Subjects with a history of allergic or anaphylactic reaction to a therapeutic drug.
* History of tuberculosis or active, latent or inadequately treated tuberculosis infection.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half lives or 180 days for biologics preceding the first dose of study medication.
* Pregnant females; breastfeeding females; and females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting or intolerability treatment related adverse events (AEs). | 6 weeks
Incidence, severity and causal relationship of treatment emergent AEs (TEAEs) and withdrawals due to treatment emergent adverse events. | 6 weeks
Incidence and magnitude of abnormal laboratory findings. | 6 weeks
Abnormal and clinically relevant changes in vital signs, blood pressure (BP) and electrocardiogram (ECG) parameters. | 6 weeks

SECONDARY OUTCOMES:
Single Ascending Dose: Maximum Observed Plasma Concentration (Cmax) | 6 weeks
Single Ascending Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) | 6 weeks
Single Ascending Dose: Area under the plasma concentration-time profile from time zero to 14 days (AUC14 days) | 6 weeks
Single Ascending Dose: Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf) | 6 weeks
Single Ascending Dose: Area under the plasma concentration-time profile from time zero to the time of last quantifiable concentration (AUClast) | 6 weeks
Single Ascending Dose: Dose normalized maximum plasma concentration (Cmax[dn]) | 6 weeks
Single Ascending Dose: Dose normalized area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf[dn]) | 6 weeks
Single Ascending Dose: Dose normalized area under the plasma concentration-time profile from time zero to the time of last quantifiable concentration (AUClast[dn]) | 6 weeks
Single Ascending Dose: Plasma Decay Half-Life (t1/2) | 6 weeks
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Single Ascending Dose: Mean residence time(MRT) | 6 weeks
Single Ascending Dose: Volume of Distribution at Steady State (Vss) | 6 weeks
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Single Ascending Dose: Systemic Clearance (CL) | 6 weeks
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Multiple Ascending Dose First Dose: Maximum Observed Plasma Concentration (Cmax) | 6 weeks
Multiple Ascending Dose First Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) | 6 weeks
Multiple Ascending Dose First Dose: Area under the plasma concentration-time profile from time zero to time τ, the dosing interval where τ=2 weeks (AUCτ) | 6 weeks
Multiple Ascending Dose First Dose: Dose normalized maximum plasma concentration (Cmax[dn]) | 6 weeks
Multiple Ascending Dose First Dose: Dose normalized Area under the plasma concentration-time profile from time zero to time τ, the dosing interval where τ=2 weeks (AUCτ [dn]) | 6 weeks
Plasma Decay Half-Life (t1/2) | 6 weeks
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Multiple Ascending Dose First Dose: Mean residence time (MRT) | 6 weeks
Apparent Volume of Distribution (Vz/F) | 6 weeks
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Multiple Ascending Dose First Dose: Volume of Distribution at Steady State (Vss) | 6 weeks
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Multiple Ascending Dose First Dose: Apparent Oral Clearance (CL/F) | 6 weeks
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Multiple Ascending Dose First Dose: Systemic Clearance (CL) | 6 weeks
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Multiple Ascending Dose Multiple Dose: Maximum Observed Plasma Concentration (Cmax) | 6 weeks
Multiple Ascending Dose Multiple Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) | 6 weeks
Multiple Ascending Dose Multiple Dose: Area under the plasma concentration-time profile from time zero to time τ, the dosing interval where τ=2 weeks (AUCτ) | 6 weeks
Multiple Ascending Dose Multiple Dose: Dose normalized maximum plasma concentration (Cmax[dn]) | 6 weeks
Multiple Ascending Dose Multiple Dose: Dose normalized Area under the plasma concentration-time profile from time zero to time τ, the dosing interval where τ=2 weeks (AUCτ [dn]) | 6 weeks
Multiple Ascending Dose Multiple Dose: Plasma Decay Half-Life (t1/2) | 6 weeks
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Multiple Ascending Dose Multiple Dose: Apparent Volume of Distribution (Vz/F) | 6 weeks
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Multiple Ascending Dose Multiple Dose: Volume of Distribution at Steady State (Vss) | 6 weeks
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Multiple Ascending Dose Multiple Dose: Apparent Oral Clearance (CL/F) | 6 weeks
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Multiple Ascending Dose Multiple Dose: Systemic Clearance (CL) | 6 weeks
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Multiple Ascending Dose Multiple Dose: Minimum Observed Plasma Trough Concentration (Cmin) | 6 weeks
Multiple Ascending Dose Multiple Dose: Average concentration at steady state (Cav) | 6 weeks
Multiple Ascending Dose Multiple Dose: Observed accumulation ratio (Rac) | 6 weeks
Multiple Ascending Dose Multiple Dose: Peak to trough fluctuation (PTF) | 6 weeks
Multiple Ascending Dose Additional Parameter: estimate of bioavailability (F) for subcutaneous administration at the corresponding intravenous dose | 6 weeks
Immunogenicity for both Single Ascending Dose and Multiple Ascending Dose: Development of anti-drug antibodies (ADA) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Banfield C, Rudin D, Bhattacharya I, Goteti K, Li G, Hassan-Zahraee M, Brown LS, Hung KE, Pawlak S, Lepsy C. First-in-human, randomized dose-escalation study of the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of PF-06480605 in healthy subjects. Br J Clin Pharmacol. 2020 Apr;86(4):812-824. doi: 10.1111/bcp.14187. Epub 2020 Jan 28. PMID 31758576
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7541001&StudyName=Study%20to%20Evaluate%20the%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20and%20Pharmacodynamics%20of%20Single%20Intravenous%20and%20Multiple%20Subcutaneous%20and%20Intr